CLINICAL TRIAL: NCT06950359
Title: Evaluation of the Effects of Cyanoacrylate and Polyglycolic Acid-Based Wound Dressings on Secondary Wound Healing
Brief Title: Comparing Two Wound Coverings for Healing and Comfort After Palatal Gum Graft Surgery in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hooman Hashemzadeh, Research Assistant, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.30.2.ODM.0.20.08/712
Record Dates: First submitted 2025-04-17; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Wound Healing
Keywords: Secondary wound healing; Periodontal surgery; Palatal wound healing; Cyanoacrylate tissue adhesive; Polyglycolic acid dressing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gelatin Sponge (Control Group) (Active Comparator): Participants (n=15) received a gelatin sponge dressing (Cutanplast®) placed over the palatal donor site and secured with crossed sling sutures around adjacent teeth.
  Interventions: Device: Gelatin Sponge Dressing (Cutanplast®)
- Cyanoacrylate Group (Test Group 1) (Experimental): Participants (n=15) received a gelatin sponge dressing (Cutanplast®), followed by application of cyanoacrylate tissue adhesive (PeriAcryl®) to the sponge and wound margins. The dressing was stabilized using crossed sling sutures.
  Interventions: Device: Gelatin Sponge Dressing (Cutanplast®); Device: Cyanoacrylate Tissue Adhesive (PeriAcryl®)
- Polyglycolic Acid Group (Test Group 2) (Experimental): Participants (n=15) received a gelatin sponge dressing (Cutanplast®) covered with a polyglycolic acid sheet (Neoveil®), trimmed to fit the wound and fixed with crossed sling sutures.
  Interventions: Device: Gelatin Sponge Dressing (Cutanplast®); Device: Polyglycolic Acid Sheet (Neoveil®)

INTERVENTIONS:
Device: Gelatin Sponge Dressing (Cutanplast®) — Absorbable gelatin-based hemostatic sponge used for all study groups as a wound contact dressing.
Device: Cyanoacrylate Tissue Adhesive (PeriAcryl®) — High-viscosity N-Butyl Cyanoacrylate/2-Octyl Cyanoacrylate adhesive applied as a topical barrier to the palatal wound site in the Cyanoacrylate Group.
  Arms: Cyanoacrylate Group (Test Group 1)
Device: Polyglycolic Acid Sheet (Neoveil®) — Bioresorbable PGA sheet placed over the gelatin sponge in the Polyglycolic Acid Group to enhance wound protection and healing.
  Arms: Polyglycolic Acid Group (Test Group 2)

SUMMARY:
After gum-grafting surgery, the bare spot in the palate can be slow to heal and quite sore. In this study, the investigators are trying three dressing methods to see which helps most: Standard care: gelatin sponge alone, Option A: gelatin sponge plus quick-dry tissue glue (cyanoacrylate), Option B: gelatin sponge plus a dissolvable mesh (polyglycolic acid). Investigators will enroll 45 adults having a free gingival graft and randomly assign 15 people to each group. Once the graft is taken, investigators will apply and suture in the assigned dressing. Follow-up visits will occur at 1 and 2 weeks, and at 1 and 2 months. Investigators will evaluate: Wound healing using two simple scales-how fast the site repairs (LTH index) and (MMS). Pain and burning sensations will also be recorded using a visual analog scale (VAS). By comparing these three approaches, investigators hope to find which dressing speeds recovery, improves the final result, and keeps discomfort to a minimum.

DETAILED DESCRIPTION:
Free gingival grafting (FGG) is a well-established periodontal procedure commonly used to increase keratinized tissue width or treat gingival recessions. However, harvesting tissue from the palate leaves a secondary wound at the donor site, which often heals by secondary intention. This can result in considerable postoperative discomfort, delayed epithelialization, and an increased risk of complications such as bleeding, infection, or scarring. This randomized, controlled clinical trial aims to compare the effectiveness of three different wound dressing approaches in promoting healing and reducing patient morbidity at the palatal donor site following FGG surgery. A total of 45 adult patients requiring FGG for periodontal or mucogingival indications will be enrolled and randomly assigned (1:1:1 ratio) into three groups: Control Group: Gelatin sponge (standard care), CYA Group (Option A): Gelatin sponge combined with a cyanoacrylate tissue adhesive (a fast-polymerizing topical glue) and PGA Group (Option B): Gelatin sponge combined with a bioresorbable polyglycolic acid (PGA) sheet. All materials used are biocompatible and approved for surgical application. After the graft is harvested, the assigned dressing will be sutured to the palatal wound under standard aseptic conditions. No additional protective stent will be used to isolate the effect of the test materials. The study is designed to evaluate and compare outcomes related to tissue healing, patient-reported pain, and wound appearance over a structured postoperative timeline. Patients will be followed up on Day 7, Day 14, and at 1 and 2 months after surgery. Objective Clinical Assessments include: Wound healing: Assessed via the Landry, Turnbull, and Howley (LTH) Index and Modified Manchester Scar Scale (MMS), Epithelialization: Measured using the hydrogen peroxide (H₂O₂) bubble test, a visual indicator of open vs. epithelialized tissue. Subjective Patient-Reported Outcomes: Pain and burning sensation: Recorded using a 0-100 Visual Analog Scale (VAS) during the first 7 postoperative days and at follow-up visits. This trial will explore whether the addition of cyanoacrylate or PGA dressing materials can improve clinical healing parameters and enhance patient comfort compared to standard gelatin sponge treatment. The hypothesis is that bioactive dressings may promote faster epithelialization and superior healing outcomes, while also minimizing early postoperative pain. The findings from this trial may contribute to developing best-practice protocols for donor site management following periodontal soft tissue grafting, with the potential to enhance recovery quality and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Good oral hygiene
* Not using any medications that affect wound healing
* No systemic diseases that may impair the normal healing process
* Non-smokers
* No clotting disorders
* Not being pregnant or in the lactation period (for female patients)

Exclusion Criteria:

* Patients with systemic conditions (e.g., diabetes, radiotherapy/chemotherapy, etc.)
* Individuals using any medication that may affect wound healing
* Individuals with coagulation disorders
* Smokers
* Pregnancy and breastfeeding
* Poor oral hygiene
* Patients who do not attend follow-up appointments regularly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
MMS (Modified Manchester Scar Scale) | Post-operative days 7, 14, and 1st month
  Healing quality assessed by scoring color, contour, and distortion. Each category: 0 (best) to 2 (worst). Total score: 0 (best) to 6 (worst).
  Scale Range: 0-6 Directionality: Lower scores = better outcome
Landry, Turnbull and Howley (LTH) healing index | Post-operative day 7, day 14, 1st month and 2nd month
  Healing quality scored from 1 (very poor) to 5 (excellent) based on redness, bleeding, granulation, epithelialization, and suppuration.
  Scale Range: 1-5 Directionality: Higher scores = better outcome
Epithelialization (H₂O₂ bubbling test) | Post-operative day 7, day 14 and 1st month
  Complete epithelialization assessed using 3% hydrogen peroxide. Positive (bubbles present) = no epithelialization Negative (no bubbles) = complete epithelialization Scale Type: Binary (Positive/Negative) Directionality: Negative result = better outcome
VAS pain score | Post-operative days 1-7, 14th day and 1st month
  Assessed using a 0-100 modified Visual Analog Scale (VAS), where 0 = no pain and 100 = worst imaginable pain. Patients recorded pain levels daily for 7 days. Additional follow-ups occurred on Day 14, and Month 1.
  Scale Range: 0-100 Directionality: Higher scores = worse outcome

SECONDARY OUTCOMES:
VAS burning sensation score | Post-operative days 1-7, 14th day and 1st month
  Assessed using a 0-100 modifed Visual Analog Scale (VAS), where 0 = no burning sensation and 100 = worst imaginable burning sensation. Patients recorded burning sensation levels daily for 7 days. Additional follow-ups occurred on Day 14, and Month 1. Scale Range: 0-100 Directionality: Higher scores = worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Hooman Hashemzadeh, DDS, Principal Investigator — Ondokuz Mayıs University; Umur Sakallıoğlu, PHD, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs Üniversitesi Diş Hekimliği Fakültesi - Ondokuz Mayis University Faculty of Dentistry, Samsun, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No